CLINICAL TRIAL: NCT06348160
Title: iHERO Study: Insurance, Health and Economic Resources Online for Emerging Adults With Type 1 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Julia Blanchette, Assistant Professor of Medicine, Nurse Scientist, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY20230187
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Health insurance; Financial stress; Young adults; Health insurance literacy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Financial Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iHERO Resource Group (Experimental): Toolkit consisting of micro-videos and supplemental online resources.
  Interventions: Behavioral: iHERO Toolkit Resource
- Control (No Intervention)

INTERVENTIONS:
Behavioral: iHERO Toolkit Resource — iHERO Toolkit consists of micro-videos and supplemental online resources. Participants will have access to the toolkit housed on pathfactory for 30 days.
  Arms: iHERO Resource Group

SUMMARY:
This research study aims to test a financial and health insurance iHERO Toolkit for young adults with type1 diabetes. The iHERO Toolkit was developed over one year with the type 1 diabetes community, The Diabetes Link organization, and experts. Now, the investigators want to understand the impact of the iHERO Toolkit on diabetes self-management, financial stress, and health insurance literacy outcomes. The investigators are doing this study because it will help to better understand how to support health insurance and financial stress and improve self-management outcomes in young adults with type 1 diabetes. The investigators want to understand how the iHERO Toolkit helps all young adults with diabetes, but especially those on Medicaid and who are racially or ethnically diverse. The investigators will ask participants to participate at four-time points over one year. For the first time, participants will fill out online enrollment and demographic forms and 9 surveys. The 9 surveys have 8-40 short questions each, estimated to take about 45 minutes. Participants will also be asked to complete a home A1c collection with a University Hospitals team member on Zoom.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-30 years
* Diagnosis of type 1 diabetes (T1D)
* T1D duration for one year or longer
* Geographical location: residing in the United States.

Exclusion Criteria:

* Inability to answer questions due to cognitive status.
* Inability to read or understand English.
* Diagnosis of insulin-dependent diabetes that is not T1D such as cystic fibrosis-related diabetes, maturity-onset diabetes of the young, or insulin-dependent type 2 diabetes.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 195 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2026-11-22 (Estimated); Study Completion 2026-11-22 (Estimated)

PRIMARY OUTCOMES:
Change in financial stress as measured by the Personal Financial Well-Being Scale© (PFW) Scale (PFW) | Baseline, 1 month, 6 months, 12 months
  The PFW is an 8-item scale used to measure financial stress with a Likert scale of 1-10 with 1 being no financial stress and 10 being an overwhelming level of financial stress. Lower scores (≤ 4.4) indicate high financial stress, while scores ranging from 4.5-6.4 indicate average stress, and scores ≥ 6.5 indicate low stress.
Change in health insurance literacy as measured by The Health Insurance Literacy Measure (HILM) Measure (HILM) | Baseline, 1 month, 6 months, 12 months
  The HILM is a 21-item measure used to rate confidence in selecting and using health insurance with 0 representing little confidence and 4 representing highest confidence. The scores of the items are summed and range from 0 to 84, with higher scores representing greater levels of health insurance literacy.
Change in diabetes-specific quality of life as measured by The Type 1 Diabetes and Life Young Adult (T1DAL- Young Adult) for ages 18-25 or The Type 1 Diabetes and Life (T1DAL- Adult) for Ages 26-30. | Baseline, 1 month, 6 months, 12 months
  T1DAL-Young Adult and T1DAL- Adult are scored on a scale of 0-100 with higher scores indicating better health related quality of life.
Change in transition navigation readiness as measured by the The Readiness for Emerging Adults with Diabetes Diagnosed in Youth (READDY) Navigation Subscale | Baseline, 1 month, 6 months, 12 months
  READDY navigation sub-scale scores of 1-3 indicate lower levels of confidence and scores of 4-5 indicate higher levels of confidence in healthcare navigation.
Change in HbA1c levels as measured by self-collect capillary HbA1c | Baseline, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Julia Blanchette, PhD, Principal Investigator — University Hospitals
Locations (4):
- United States (4):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Florida Diabetes Institute, Gainesville, Florida
  - University Hospitals, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanchette JE, Toly VB, Wood JR. Financial stress in emerging adults with type 1 diabetes in the United States. Pediatr Diabetes. 2021 Aug;22(5):807-815. doi: 10.1111/pedi.13216. Epub 2021 May 18. PMID 33887095
- [Background] Blanchette JE, Allen NA, Litchman ML. The Feasibility and Acceptability of a Community-Developed Health Insurance and Financial Toolkit for Emerging Adults With Type 1 Diabetes. Sci Diabetes Self Manag Care. 2022 Jun;48(3):174-183. doi: 10.1177/26350106221087474. Epub 2022 Mar 15. PMID 35287511